CLINICAL TRIAL: NCT05330650
Title: Evaluation of Triclosan Coated Suture in Obstetrical Surgery: A Randomized Controlled Study
Brief Title: Evaluation of Triclosan Coated Suture in Obstetrical Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tunis University (Other)
Responsible Party: Principal Investigator, Hajer BETTAIEB, Assistant professor, Tunis University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TunisU 1
Record Dates: First submitted 2022-03-21; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Cesarean Section; Infection
Keywords: Surgical Site Infections; caesarean section; healthcare costs
MeSH Terms: conditions — Infections; Surgical Wound Infection | interventions — Polyglactin 910

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triclosan coated suture (Active Comparator)
  Interventions: Drug: Coated Vicryl+
- Non coated suture (Active Comparator)
  Interventions: Drug: Vicryl

INTERVENTIONS:
Drug: Coated Vicryl+ — We used coated suture for : hystetrotomy reparation / aponeurosis and skin closure.
  Arms: Triclosan coated suture
Drug: Vicryl — We used non coated suture for : hystetrotomy reparation / aponeurosis and skin closure.
  Arms: Non coated suture

SUMMARY:
A prospective comparative randomized blinded study conducted in the obstetrics gynecology department of Ben Arous hospital over an eight-month period between November 2020 and June 2021.

The aim of this study is to evaluate effectiveness of Triclosan coated suture use in obstetrical surgery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with indicated cesarean delivery and who have signed a written consent.

Exclusion Criteria:

* Cases with incomplete follow up
* Breach of operative protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of surgical site infection | 30 days

SECONDARY OUTCOMES:
Health care costs attributable to surgical site infection | 30 days
  Evaluation of health care costs from Hospital perspective (USD)
Wound healing time | 30 days
  Evaluation of healing time (days)

CONTACTS AND LOCATIONS:
Overall Officials: Chaouki Mbarki, Study Director — Ben Arous Hospital, Tunis, Tunisia
Locations (1):
- Obstetrics and Gynecology Departement, Ben Arous, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mbarki W, Bettaieb H, Souayeh N, Laabidi I, Rouis H, Halouani S, Boufarghine R, Bouyahia M, Bouhmida R, Ouederni M, Ben Amor A, Chermiti A, Laamiri H, Lika A, Chaibi I, Oueslati H, Hsayaoui N, Mbarki C. Evaluation of Triclosan coated suture in obstetrical surgery: A prospective randomized controlled study (NCT05330650). PLoS One. 2022 Dec 15;17(12):e0278939. doi: 10.1371/journal.pone.0278939. eCollection 2022. PMID 36520813